CLINICAL TRIAL: NCT03625596
Title: The Effects of Nutritional Supplements on Postprandial Nitric Oxide Bioactivity in Abdominally Obese Men
Brief Title: Nutritional Supplements and Nitric Oxide Bioactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 18-3-010
Record Dates: First submitted 2018-07-24; First posted 2018-08-10 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Nitric Oxide; Vascular Function; L-Arginine; Nitrate / Nitrite; Postprandial Metabolism
MeSH Terms: interventions — Arginine; Nitrates; Nitrites

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- High L-arginine (Active Comparator): During this experimental day, men will receive a high-fat shake with a high dose of L-arginine.
  Interventions: Dietary Supplement: L-Arginine
- Medium L-arginine + Nitrate / Nitrite (Experimental): During this experimental day, men will receive a high-fat shake with a medium dose of L-arginine enriched with nitrate and nitrite.
  Interventions: Dietary Supplement: L-Arginine; Dietary Supplement: Nitrate / Nitrite
- Low L-arginine + Nitrate / Nitrite (Experimental): During this experimental day, men will receive a high-fat shake with a low dose of L-arginine enriched with nitrate and nitrite.
  Interventions: Dietary Supplement: L-Arginine; Dietary Supplement: Nitrate / Nitrite
- Nitrate / Nitrite (Experimental): During this experimental day, men will receive a high-fat shake with nitrate and nitrite.
  Interventions: Dietary Supplement: Nitrate / Nitrite
- Placebo (Placebo Comparator): During this experimental day, men will receive a high-fat shake without supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Arginine — Acute intervention (3 hours)
  Arms: High L-arginine; Low L-arginine + Nitrate / Nitrite; Medium L-arginine + Nitrate / Nitrite
Dietary Supplement: Nitrate / Nitrite — Acute intervention (3 hours)
  Arms: Low L-arginine + Nitrate / Nitrite; Medium L-arginine + Nitrate / Nitrite; Nitrate / Nitrite
Dietary Supplement: Placebo — Acute intervention (3 hours)
  Arms: Placebo

SUMMARY:
Obese people have a disturbed postprandial metabolism and thereby a decreased postprandial vascular function. Nitric oxide plays an important role in the postprandial vascular function. Multiple studies already focused on various nutritional compounds to improve the postprandial vascular function by increasing the nitric oxide bioactivity. However, the vast majority of the trials has been performed with relatively high doses of the individual components, which are problematic to convert into daily food measures, thereby preventing translation of these findings. Well-designed trails studying the effect of feasible amounts of nutritional supplements on the bioactivity of nitric oxide and vascular function are missing.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Aged between 40-70 years
* Waist circumference ≥ 102
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* No more than 3 alcoholic consumptions per day
* No use of medication known to treat blood pressure, lipid or glucose metabolism
* No use of an investigational product within another biomedical intervention trial within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Willingness to give up the use of antibacterial mouth wash or antibacterial toothpaste, chewing-gum and tongue- scraping on the morning of each experimental test day

Exclusion Criteria:

* Women
* Fasting plasma glucose ≥ 7.0 mmol/L
* Fasting serum total cholesterol ≥ 8.0 mmol/L
* Current smoker, or smoking cessation <12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use medication known to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Nitric oxide bioavailability | Change from baseline at 2 hours after supplement intake
  Flow-mediated vasodilation (FMD) of the brachial artery

SECONDARY OUTCOMES:
Nitric oxide bioavailability | During 3 hours following supplement intake
  Plasma cyclic guanosine monophosphate (cGMP)
Vascular function markers | Change from baseline at 2 hours after supplement intake
  Retinal microvascular calibers
Cardiometabolic risk markers (1) | Change from baseline at 2 hours after supplement intake
  Plasma markers for low-grade systemic inflammation (CRP)
Cardiometabolic risk markers (2) | Change from baseline at 2 hours after supplement intake
  Plasma markers for endothelial dysfunction (NOx)
Cardiometabolic risk markers (3) | Change from baseline at 2 hours after supplement intake
  Office blood pressure
Postprandial metabolism (1) | During 3 hours following supplement intake
  Serum lipid metabolism
Postprandial metabolism (2) | During 3 hours following supplement intake
  Plasma glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands